CLINICAL TRIAL: NCT05658003
Title: An Open-label, Multi-center, Randomized, Phase II Study Evaluating [177Lu]Lu-PSMA-617 vs. a Change of Androgen Receptor-directed Therapy in the Treatment of Taxane Naive Chinese Male Patients With Progressive Metastatic Castrate Resistant Prostate Cancer
Brief Title: A Study Evaluating [177Lu]Lu-PSMA-617 vs. a Change of Androgen Receptor-directed Therapy in Taxane Treatment Naive Chinese Male Patients With Progressive Metastatic Castrate Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAA617B12201
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Chinese adult male population; therapeutic agent lutetium (177Lu) vipivotide tetraxetan; [177Lu]Lu-PSMA-617; Progressive PSMA-Positive Metastatic Castration-Resistant Prostate Cancer; rPFS; Prostate-specific Membrane Antigen; PSMA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [177Lu]Lu-PSMA-617 (Experimental): Participants will receive 7.4 GBq (200 mCi) +/- 10% [177Lu]Lu-PSMA-617 once every 6 weeks for 6 cycles. Best supportive care, including ADT may be used.
  Interventions: Drug: [177Lu]Lu-PSMA-617; Drug: [68Ga]Ga-PSMA-11; Other: Best supportive care
- Androgen receptor-directed therapy (ARDT) (Active Comparator): For participants randomized to the ARDT arm, the change of ARDT treatment will be administered per the physician's orders. Best supportive care, including ADT may be used.
  Interventions: Drug: ARDT; Drug: [68Ga]Ga-PSMA-11; Other: Best supportive care

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA-617 — administered intravenously once every 6 weeks (1 cycle) for 6 cycles
  Arms: [177Lu]Lu-PSMA-617
Drug: ARDT — administered orally on a continuous basis, as per package insert and guidelines
  Other Names: Comparator
  Arms: Androgen receptor-directed therapy (ARDT)
Drug: [68Ga]Ga-PSMA-11 — single intravenous dose of approximately 150 MBq. Administered dose must not be lower than 111 MBq or higher than 259 MBq (3 - 7 mCi).
Other: Best supportive care — Best supportive/best standard of care as defined by the local investigator

SUMMARY:
The purpose of this study is to evaluate the efficacy of [177Lu]Lu-PSMA-617 over a change of androgen receptor-directed therapy (ARDT) treatment in prolonging radiographic progression free survival (rPFS) in Chinese metastatic castration-resistant prostate cancer patients, who were previously treated with another ARDT as last treatment and who have not been exposed to a taxane-containing regimen in castrate resistant prostate cancer (CRPC) or hormone-sensitive prostate cancer (HSPC) settings and who are considered appropriate for delaying taxane-based chemotherapy. The primary endpoint of rPFS will be assessed via blinded independent centralized review of radiographic images provided by the treating physician and as outlined in Prostate Cancer Working Group 3 (PCWG3) guidelines.

DETAILED DESCRIPTION:
The study contains a screening period to assess the eligibility of participants, only participants fulfilling the [68Ga]Ga-PSMA-11 PET scan interpretation criteria for eligibility and meeting all other inclusion/exclusion criteria will be enrolled. In the randomization period, approximately 60 participants will be randomized 1:1 to receive [177Lu]Lu-PSMA-617 treatment or a change of approved ARDT treatment. Randomization will be stratified by symptomatology i.e., Asymptomatic or mildly symptomatic vs. symptomatic.

Participants randomized to [177Lu]Lu-PSMA-617 treatment group will receive 7.4 GBq (200 mCi) ± 10% [177Lu]Lu-PSMA-617 once every 6 weeks (± 1 week) for 6 cycles. For participants randomized to the ARDT treatment arm, the change of ARDT treatment for each participant will be selected by the treating physician prior to randomization and will be administered per the physician's orders. Supportive care will be allowed in both arms at the discretion of the investigator. ARDT must not be administrated concomitantly with [177Lu]Lu-PSMA-617.

Efficacy assessment will be performed every 8 weeks after first dose of study treatment for the first 24 weeks (week 9, 17, 25) and then every 12 weeks (week 37, 49, etc) until confirmation of radiographic progression by BICR. Upon confirmation of rPFS by BIRC, participants randomized to ARDT arm will be allowed to crossover to [177Lu]Lu-PSMA-617 treatment if the crossover criteria are met. Post-treatment follow up period will have a 30-day safety follow up post EOT visit and long term survival follow up.

ELIGIBILITY:
Key Inclusion criteria

1. Participants must be Chinese adult men >= 18 years of age
2. Participants must have an ECOG performance status of 0 to 1
3. Participant must have histological pathological and/or cytological confirmation of adenocarcinoma of the prostate
4. Participants must be [68Ga]Ga-PSMA-11 PET/CT scan positive, and eligible as determined by the sponsor's central reader
5. Participants must have a castrate level of serum/plasma testosterone (< 50 ng/dl, or < 1.7 nmol/L)
6. Participants must have progressed only once on prior second generation ARDT (abiraterone, enzalutamide, darolutamide, or apalutamide)) in either HSPC or CRPC setting.

   * first generation androgen receptor inhibitor therapy (e.g. bicalutamide) is allowed but not considered as prior ARDT therapy
   * second generation ARDT must be the most recent therapy received
7. candidates for change in ARDT (eligible to receive abiraterone or enzalutamide) as assessed by the treating physician

   • Participants cannot have previously progressed nor had intolerable toxicity to both enzalutamide and abiraterone
8. Documented progressive mCRPC, based on at least 1 of the following criteria:

   * Serum/plasma PSA progression defined as 2 consecutive increases in PSA measured at least 1 week apart. the minimal start value is 2.0 ng/ml;
   * Soft-tissue progression defined based on PCWG3-modified RECIST v1.1(Eisenhauer et al 2009, Scher et al 2016)
   * Progression of bone disease: two new lesions; only positivity on the bone scan defines metastatic disease to bone (PCWG3 criteria Scher et al 2016)
9. Participants must have at least one metastatic lesion that is present on screening/baseline CT, MRI, or bone scan imaging obtained =< 28 days prior to randomization
10. Participants must have adequate organ function:

    * Bone marrow reserve:
    * ANC >= 1.5 x 109/L
    * Platelets >= 100 x 109/L
    * Hemoglobin >= 9 g/dL
    * Hepatic:
    * Total bilirubin < 2 x the institutional upper limit of normal (ULN). For participants with known Gilbert's Syndrome =< 3 x ULN is permitted
    * ALT or AST =< 3.0 x ULN OR =< 5.0 x ULN for participants with liver metastases
    * Albumin >= 2.5 g/dL
    * Renal:
    * eGFR >= 50 mL/min/1.73m2 using the Modification of Diet in Renal Disease (MDRD) equation

Key Exclusion criteria

1. Previous treatment with any of the following within 6 months of randomization: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, Lutitium-177, Actium-225, hemi-body irradiation
2. Previous PSMA-targeted radioligand therapy
3. Prior treatment with PARP inhibitor, cytotoxic chemotherapy for castration resistant or castration sensitive prostate cancer (i.e., taxanes, platinum, estramustine, vincristine, methotrexate, etc.), immunotherapy or biological therapy (including monoclonal antibodies). [Note: a maximum of 6 cycles of taxane exposure in the adjuvant or neo-adjuvant setting is allowed if 12 months have elapsed since completion of this adjuvant or neo-adjuvant therapy prior to randomization]
4. Concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, PARP inhibitor, biological, or investigational therapy
5. Transfusion or use of bone marrow stimulating agents for the sole purpose of making a participant eligible for study inclusion
6. Participants with a history of CNS metastases who are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity.

   * Participants with CNS metastases are eligible if received therapy (surgery, radiotherapy, gamma knife), asymptomatic and neurologically stable without corticosteroids.
   * Participants with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired.
7. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression
8. Cardiac or cardiac repolarization abnormality, including any of the following:

   * History of myocardial infarction (MI), angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to starting study treatment
   * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block) and QTc>=500.
9. Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, known active hepatitis B or C or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation
10. Unmanageable concurrent bladder outflow obstruction or urinary incontinence. Note: Participants with bladder outflow obstruction or urinary incontinence, which is manageable and controlled with best available standard of care (incl. pads, drainage) are allowed.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 62 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2027-01-13 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression free survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 42 months
  Radiographic progression free survival (rPFS) is defined as the time of radiographic progression by Prostate Cancer Working Group 3 (PCWG3)-modified RECIST V1.1 as assessed by blinded independent central review, or death.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until date of death from any cause, assessed up to 59 months (estimated final OS analysis)
  Overall survival (OS) is defined as the time from the date of enrollment to the date of death due to any cause. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive (on or before the cut-off date).
Progression Free Survival (PFS) | From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up to 59 months (estimated final OS analysis)
  Progression Free Survival (PFS) is defined as the time from date of randomization to the date of first documented progression by investigator assessment (radiographic progression, clinical progression, PSA progression) or death from any cause, whichever occurs first.
Prostate-specific antigen 50 response rate | Week 12, Week 24, Week 48
  PSA 50 response rate is the proportion of PSA responders, defined as a participant who has achieved PSA decrease of >= 50% from baseline that is confirmed by a second consecutive PSA measurement >= 4 weeks later. Determination of response status will be based on PCWG3 recommendations.
Time to a first symptomatic skeletal event (TTSSE) | From date of randomization till date of death from any cause, whichever happens first, assessed up to 59 months (estimated final OS analysis)
  Time to a first symptomatic skeletal event (TTSSE) is defined as date of randomization to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first.
Time to Prostate Specific Antigen (PSA) progression | From date of randomization till date of Prostate Specific Antigen (PSA) progression, assessed up to 59 months (estimated OS analysis)
  Time to PSA Progression (TTPSAP) defined as time from randomization to PSA progression. PSA progression date is defined as the date of 1) >= 25% increase and >= 2 ng/mL above the nadir, confirmed by a second value >= 3 weeks later if there is a PSA decline from baseline, or 2) >= 25% increase and >= 2ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline:
Time to chemotherapy (TTCT) | From date of randomization until date of subsequent chemotherapy or date of death from any cause, whichever comes first, assessed up to 59 months (estimated final OS analysis)
  Time to chemotherapy (TTCT) defined as time from randomization to initiation of the first subsequent chemotherapy or death, whichever occurs first.
Overall response rate (ORR) | From date of randomization till 30 day safety follow-up or end of long term FU for patients prematurely discontinued, assessed up to 59 months (estimated final OS analysis)
  Overall response rate (ORR)is defined as the proportion of participants with best overall response of complete response or partial response in soft tissue as per BIRC and according to PCWG3 modified RECIST 1.1
Disease control rate (DCR) | From date of randomization till 30 day safety follow-up or end of long term FU for patients prematurely discontinued, assessed up to 59 months (estimated final OS analysis)
  Disease control rate (DCR) is defined as the proportion of participants with best overall response of complete response or partial response or Stable disease in soft tissue as per BIRC and according to PCWG3 modified RECIST 1.1
Time to response (TTR) | From date of randomization till 30 day safety follow-up or end of long term FU for patients prematurely discontinued, assessed up to 59 months (estimated final OS analysis)
  Time to response (TTR) is defined as the time from the date of randomization to the date of first documented response (CR or PR, which must be confirmed subsequently). CR and PR are based on tumor response data as per BICR and according to PCWG3-modified RECIST v1.1. Participants who did not achieve a confirmed CR or PR will be censored at the last adequate tumor assessment date when they did not have a PFS event or at maximum follow-up (i.e. FPFV to LPLV used for the analysis) when they did have a PFS event.
Duration of response (DOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 59 months (estimated final OS analysis)
  Duration of response (DOR) is defined as the duration of time between the date of first documented response (CR or PR) in soft tissue as per BIRC and according to PCWG3 modified RECIST 1.1, and the date of first documented progression or death due to any cause.
Time to soft tissue progression (TTSTP) | From date of randomization until date of soft tissue radiographic progression or date of death from any cause, whichever comes first, assessed up to 59 months (estimated final OS analysis)
  Time to soft tissue progression (TTSTP) defined as time from randomization to radiographic soft tissue progression per PCWG3-modified RECIST v1.1 assessed by BICR.
European Quality of Life (EuroQol) - 5 Domain 5 Level scale (EQ-5D- 5L) | From randomization up till 30 day safety follow-up or at LTFU2 (168 days after EOT) and LTFU4 (336 days after EOT) of long term FU for patients prematurely discontinued, assessed up to 59 Months (estimated final OS analysis)
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire | From randomization up till 30 day safety follow-up or at LTFU2 (168 days after EOT) and LTFU4 (336 days after EOT) of long term FU for patients prematurely discontinued, assessed up to 59 Months (estimated final OS analysis)
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Brief Pain Inventory - Short Form (BPI-SF) Questionnaire | From randomization up till 30 day safety follow-up or at LTFU2 (168 days after EOT) and LTFU4 (336 days after EOT) of long term FU for patients prematurely discontinued, assessed up to 59 Months (estimated final OS analysis)
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
Number of Participants with Treatment Emergent Adverse Events | From date of randomization till 30 days safety fup, assessed up to 59 months (estimated final OS analysis)
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs), through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- China (10):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com